Dear Sir or Madam:

We are conducting a study to investigate the effects of postures on time up and go. In this study, we will measure the time is required for you to stand up from a chair, walk for 10 feet, and return to sit down in the chair. We will take the aforementioned baseline measurements first, and then we will ask you to hold a certain posture for 20 seconds. Immediately after you have held the posture for 20 seconds, we will take the measurements again. We will also need to collect information to describe you such as age or gender. You will meet with us for one session and your participation should take about ten minutes.

Standing for 20 seconds poses a minimal risk to you. The outcome measurement is routinely used in physical therapy practice. To our knowledge, there are no risks or other adverse events associated with these practices. The likelihood that you will be harmed is minimized because we will monitor all physical discomfort throughout the study and no personal identifying information will be collected that could be connected to your personal results.

There are no direct benefits to participate in this study. Benefits to society include the advancement of scientific knowledge for the profession of physical therapy by improving patient outcomes.

Your privacy is important and we will handle all information collected about you in a confidential manner. We will report the results of the project in a way that will not identify you. We plan to submit the results to professional conference presentation and journal publication.

You do not have to be in this study. If you don't want to, you can say no without any negative consequences. If you do agree, you can stop participating at any time. If you wish to withdraw just tell us or the contact person listed below.

If you have questions about this research project please contact Weiqing Ge, DPT, PhD, Associate Professor of Physical Therapy at (330) 941-2702. If you have questions about your rights as a participant in a research project, you may contact the Office of Research at YSU (330-941-2377) or at YSUIRB@ysu.edu.

| If the participant is of age (18 years old I understand the study described above a years of age or older and I agree to partic | nd have been given a copy of t | his consent document. I am 18 |
|---|---|---|
| Signature of Participant | Date | |